CLINICAL TRIAL: NCT02486419
Title: Human Neck Brown Adipose Tissue mRNA Profile, a Seasonal Variation Study.
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Peter Breining, MD PhD student, Aarhus University Hospital
Other Study IDs: 1-10-72-297-14
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Nonshivering Thermogenisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Adipose tissue biopsies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Summer
  Interventions: Other: Outdoor weather
- Winter
  Interventions: Other: Outdoor weather

INTERVENTIONS:
Other: Outdoor weather — Seasonal changes in temperature

SUMMARY:
The primary objective in this study is to examine the seasonal variation in genetic markers in the deep neck adipose tissue in humans.

Human adipose tissue biopsies are taken from patients admitted for elective surgery in the neck. During the surgical procedure a subcutaneous adipose tissue biopsy is taken for reference.

DETAILED DESCRIPTION:
The knowledge of brown adipose tissue (BAT) is derived mainly from studies in rodents where cold is an important regulator of BAT development and function. Yet, little is known about the regulation of BAT in humans.

With this study the investigators aim to investigate the effects of seasonal changes in outdoor temperature on genetic markers of BAT in human deep neck adipose tissue.

Project participants are patients who are admitted to Aarhus University Hospital for elective neck surgery. Operations are primarily due to suspected malignancy in the thyroid gland or hyperparathyroidism.No additional surgery is necessary to obtain the biopsies.

ELIGIBILITY:
Inclusion Criteria:

* written concent

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted for neck surgery at Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Differences in gene expression in BAT associated genes (PGC1a, UCP1, CIDEA, PRDM16) | 1 day (The biopsies will be taken as a "point in time" value. Differences between seasons will be assesed. And so will correlations between genes at one point in time.)
  biopsies will be grouped depending on outdoor temperature, differences in subcutaneous- and deep neck values,

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Richelsen, MD, PhD, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark